| Study Title: The Effect of Productivity Training on Perceived Job Stress and Productivity Attitudes in Nurses: A Randomized Controlled Experimental Study |
|---|
| ClinicalTrials.gov Identifier: Not yet assigned |
| Document Type: Informed Consent Form |
| Date: 11 June 2025 |

## INFORMED CONSENT FORM

You are invited to participate in a research study entitled "The Effect of Productivity Training on Perceived Job Stress and Productivity Attitudes in Nurses: A Randomized Controlled Experimental Study", conducted by MSc student Neslihan Erim under the supervision of Dr. Seyhan Çerçi at Istanbul Arel University Graduate Education Institute.

The purpose of this study is to evaluate nurses' productivity-related attitudes and perceived job stress levels. If you agree to participate, you will be asked to complete the data collection forms, which will take approximately **5 minutes**.

Participation in this study is entirely voluntary. You have the right to refuse participation or to withdraw from the study at any time without any penalty or negative consequences. No payment will be made to you for participating in this study, and no costs will be incurred.

All information collected in this study will be used solely for research purposes. Your personal information will be kept confidential and anonymous. The data obtained may be used for scientific publications; however, your identity will not be disclosed.

By completing the questionnaire, you indicate that you have read and understood the information provided above and voluntarily agree to participate in this study. You acknowledge that you may withdraw from the study at any time without any consequences.

Thank you very much for your participation and for taking the time to contribute to this research.

## Researcher:

Neslihan Erim, RN

## **Supervisor:**

Dr. Seyhan Çerçi